CLINICAL TRIAL: NCT07273305
Title: Effect of Cultural Competence Training on Nurses' Cultural Competence Levels and Patients' Perceptions of Culturally Competent Care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oyku Ozturk (Other)
Responsible Party: Sponsor-Investigator, Oyku Ozturk, PhD Candidate, Clinical Research Nurse, Koç University
Organization: Koç University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: KUN-OO-001
Record Dates: First submitted 2025-11-26; First posted 2025-12-09 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Cultural Competence Training in Nursing

STUDY DESIGN:
Intervention Model Description: Two-group randomized pretest-posttest parallel design comparing the effect of cultural competence training on nurses' cultural competence levels and patient perceptions.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): The nurse who is in intervention arm will be in training programme.
  Interventions: Behavioral: Cultural Competence Training Program
- Control Arm (No Intervention): The nurse in the control group will not undergo any procedure.

INTERVENTIONS:
Behavioral: Cultural Competence Training Program — A four-week behavioral educational program designed to improve nurses' cultural competence, based on Tanrıverdi's Environment-Oriented Cultural Competence Model. The program involves interactive lectures, case discussions, and reflection-based exercises focused on culturally competent care practices. Educational program is still developing, so it can be changed.
  Arms: Intervention Arm

SUMMARY:
This study aims to evaluate the effectiveness of a cultural competence training program based on Gülbu Tanrıverdi's Environment-Oriented Cultural Competence Model in improving nurses' cultural competence levels and in enhancing patients' perceptions of culturally competent care. The study adopts a mixed-method design including a randomized controlled pre-test/post-test intervention for nurses and semi-structured interviews with patients from diverse cultural backgrounds.

ELIGIBILITY:
Inclusion Criteria:

* Have not previously received any training on transcultural nursing or cultural competence

Currently working in units that provide care to international adult patients

Not holding a managerial or administrative position

Voluntarily agree to participate in the study

Exclusion Criteria:

* Have lived or stayed abroad for more than six months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-07 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change in Nurses' Cultural Competence Score | Baseline (Pre-test, Week 0) and after completion of the 4-week training (Post-test, Week 4)
  The primary outcome will be the change in nurses' cultural competence levels before and after the training intervention. Cultural competence will be measured using the Nurse Cultural Competence Scale (NCCS), which assesses awareness, knowledge, sensitivity, and skills related to culturally competent care.

CONTACTS AND LOCATIONS:
Locations (1):
- Koc University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The individual-level data will not be shared outside the research team. Only aggregated and anonymized results will be published in academic journals.